CLINICAL TRIAL: NCT04602559
Title: Exploratory Study to Evaluate the Clinical Benefits of Wearing the Panty MOBIDERM in Patients With Pelvic and/or Genital Lymphedema : OLYMPY Study
Brief Title: Exploratory Study : to Evaluate the Panty MOBIDERM in Patients With Pelvic and/or Genital Lymphedema
Acronym: OLYMPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC31; ANSM (Other: 2020-A00247-32)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Lymphedema of Genitalia
Keywords: genital lymphedema; panty; compression; volume reduction; quality of life; pelvic lymphedema

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, interventional, open-label, prospective exploratory study in a population of patients with primary or secondary pelvic and/or genital lymphedema
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOBIDERM Panty group (Experimental): MOBIDERM Panty group :
  All patients will wear the Panty MOBIDERM device for 12 weeks, day and night recommended. A removable pad is also recommended to be worn additionnaly to the panty.
  Interventions: Device: MOBIDERM Panty group

INTERVENTIONS:
Device: MOBIDERM Panty group — In the MOBIDERM Panty group, patients wear the MOBIDERM Panty during day and night for 3 months with the possibility to add the PAD.
  The protocol includes 3 visits.
  Visit 1 at day 0, corresponding to the inclusion visit, includes device delivery and some clinical evaluations (clinical examination, characteristics of lymphedema, self questionnaires, pain assessment, perimeter data).
  Visit 2 at 30 days after the inclusion : includes some clinical evaluations (clinical examination, characteristics and evolution of lymphedema, self questionnaires, pain assessment, perimeter data, safety, compliance).
  Visit 3 at 90 days after the inclusion : includes some clinical evaluations (clinical examination, characteristics and evolution of lymphedema, self questionnaires, pain assessment, perimeter data, safety, compliance).

SUMMARY:
Lymphedema (LO) is a chronic and disabling condition that affects quality of life. This pathology has a physical, psychological, social and professional impact. Pelvic or genital lymphedema (LP/LG) is the result of a dysfunction of the lymphatic system in the genital area that can occur following surgery, radiation therapy, tumor, infections affecting the inguinal lymph nodes or related lymphatic pathways (secondary LP/LG). Urogenital cancers are the major cause of secondary LP/LG. It is difficult to have an accurate estimate of the prevalence of LP/LG. LP/LG can be painful, the edema very bulky and disharmonious. The patient is facing with significant physical and psychological difficulties. The volume of the lymphedema can be important, causing discomfort, rubbing when walking or during physical activities, disrupting daily life and may constitute a major handicap.

DETAILED DESCRIPTION:
Currently, there is no reference treatment which is validated for these lymphedemas, and few recommendations from the competent authorities or learned societies are available. There is no solution available on the market which covers all the needs and expectations of patients and healthcare professionals.

The Panty MOBIDERM is a standard pelvic compressive orthosis that should promote lymphatic drainage, then reduce the volume of edema, and contributing to an overall improvement in the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary pelvic or genital lymphedema of stage II ou III according to the criteria defined by the International Society of Lymphology.
* Patient with discomfort related to lymphedema
* Presence of the Stemmer's sign if applicable
* Patient with a morphology compatible with the 6 sizes of the MOBIDERM Panty (Minimum and maximum pelvic circumference: 88 and 129 cm respectively)
* Patient who gave signed, informed, voluntary consent prior to any intervention in the study
* Patient affiliated to the General regime of the Social Security or covered by a similar health insurance system

Exclusion Criteria:

* Pregnant woman or woman of childbearing age without contraception
* Patient with surgery of the small pelvis or genitals performed within the last 3 months prior to inclusion or any surgery scheduled during the study period
* Patient with hydrocoele
* Patient who had intensive reduction therapy for lower limb lymphedema within the last month
* Patient with a contraindication to compression, such as untreated infection, skin irritation, recent thrombosis (< 3 months), obliterative arterial disease of the lower limbs with a systolic pressure index < 0.6, phlegmatia coerulea dolens (painful blue phlebitis with arterial compression) in the thigh area
* Patient with decompensated heart failure
* Patient with a known allergy to the components used in the Panty
* Patient with untreated or escaped cancer
* Patient with a postectomy within the last 3 months prior to inclusion
* Patient with significant edema localized only to the labia minora
* Patient with psychiatric, psychological or neurological disorders that are incompatible with proper follow-up of a clinical study
* Patient participating in other research involving the human person impacting the main judgement criteria
* Patient cannot be followed for 12 weeks
* Vulnerable patient according to article L1121-6 of the French public health code, or subject being the object of a legal protective measure or enable to express his consent freely

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL): Patient's opinion on Global Impression of Change (PGI-C) | 90 days
  The patient's impression of overall change is measured by the Patient's opinion on Global Impression of Change questionnaire. The scale has 7 levels of response :
  "no change or condition has got worse" that is the worst outcome (= 1 point) "almost the same, hardly any change at all" (= 2 points); "a little better , but no noticeable change" (= 3 points); "somewhat better, but the change has not made any real difference" (= 4 points); "moderately better, and a slight but noticeable change" (= 5 points); "better, and a definite improvement that has made a real and worthwhile difference (=6 points) "A great deal better, and a considerable improvement that has made all the diiference" (=7 points) The highest score corresponds to the most improvement in quality of life.

SECONDARY OUTCOMES:
Quality of life (QoL): Lymphedema Quality of Life Inventory (LyQLI) self-questionnaire | day : 0, 30, 90
  The evolution of quality of life is measured by the lymphedema Quality of life Inventory self-questionnaire. This tool is designed as a patient-completed questionnaire.
  It comprises 45 items. Forty-one items are divided into three multi-item domains: physical (12 questions), psychosocial (16 questions), and practical (13 questions).
  For each item, the impact of lymphedema over the last 4 weeks is assessed on a 4-point Likert scale (0: None, 1: A little bit, 2: Somewhat, 3: A lot). Scores are presented as the mean for each domain, ranging from 0.0 to 3.0. A higher score indicates lower QoL. The questionnaire also includes four global questions, of which item 44 assesses the overall experience of lymphedema and item 45 the overall quality of life, both on a 4-point Likert scale ranging from 0:Very bad to 3: Very good. A higher score indicates higher QoL.
Swelling, tension, discomfort and feeling of heaviness :Visual Analog Scale (VAS) | day : 0, 30, 90
  Evolution of swelling, tension, discomfort, feeling of heaviness are measured by a visual analog scale : 0 corresponds to no discomfort/no problem (better outcome) and 10 to maximum discomfort/maximum problem (worst outcome)
Impact of lymphedema on sexual life : Visual Analog Scale (VAS) | day : 0, 30, 90
  The impact of lymphedema on patients sexual life is measured by a visual analog scale : 0 corresponds to no discomfort (better outcome) and 10 to maximum discomfort preventing sexual relation (worst outcome)
Pain : Visual Analog Scale (VAS) | day : 0, 30, 90
  Evolution of pain is measured by VAS : 0 corresponds to no pain and 10 to the maximum pain.
Sleep quality : Jenkins self-questionnaire | day : 0, 30, 90
  The evolution of sleep quality is measured by Jenkins self-questionnaire. This scale is composed of four questions about the quality of sleep.
  Each answer is scored from 0 to 5 (0=none; 1= 1-3 days; 2 = 4-7 days; 3 = 8-14 days; 4 = 15-21 days; 5 = 22-31 days) A higher score corresponds to a bad quality of sleep.
Doctors' opinion on the change of patient's health condition (Clinical Global Impression -Improvement) | day : 30, 90
  Doctors' opinion on the change of patient's health condition due to lymphedema is measured by the Clinical Global Impression - Improvement questionnaire. The scale has 7 levels of answer from "very strongly improved" which is the better outcome (= 1 point) to "very strongly aggravated" which is the worst outcome (= 7 points) .Intermediate levels are: " Significantly improved "(= 2 points) ; " Slightly improved " (= 3 points) ; " No improvement " (=4 points) ; " Slightly worsen " (=5 points) ; " Seriously worsen" ( = 6 points).
  The highest score corresponds to the most impairment in quality of life.
Characteristic of pelvic lymphedema : Genital Lymphedema Score (GLS) | day : 0, 30, 90
  The evolution of pelvic lymphedema characteristics is measured by GLS questionnaire including different fields (feeling of heaviness, feeling of tension, swelling, urinary disorders, lymphatic papillomatosis, genital lymphorrhea), and by taking pictures.
  (0= absence of the symptom,1 or 2 = presence of the symptom)
Pelvic/genital lymphedema perimetry for men only : Whitaker tool | day : 0, 30, 90
  The evolution of the pelvic/genital lymphedema is measured by perimetric measurements according to the Whitaker tool :
  Measure A: middle of the scrotum Measure B: scrotal neck size Measure C: length of the scrotum
Day and NIght Compliance to treatment | day : 30,90
  Compliance to treatment is reported by the physician in the electronic Case Report Forms (eCRF) according to the patient diary. The compliance is measured by calculating the number of days and nights corresponding to a wearing of the device The average wearing time is : Full day/night, >50% of the day/night,<50% of the day/night, not at all
Satisfaction about the device: specific self questionnaire | Day : 30
  Patient's and doctor's satisfaction with regards to MOBIDERM Panty by a satisfaction questionnaire. This questionnaire is focused on the product positioning and the comfort.
  These are qualitative variables; there is no score.
Safety: Adverse Device Effects | day : 0, 30, 90
  Number and type of serious and non-serious Adverse Device Effects (ADE) are reported all along the study.
Quality of life (QoL): EQ-5D-5L questionnaire | day : 0, 30, 90
  The evolution of quality of life is measured by the EQ-5D-5L questionnaire. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (Level 1 is coded as a '1'), slight problems (Level 2 is coded as a '2'), moderate problems (Level 3 is coded as a '3'), severe problems (Level 4 is coded as a '4'), and extreme problems (Level 5 is coded as a '5'). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS is measured by VAS : 100 corresponds to the best health and 0 to the the worst health.

CONTACTS AND LOCATIONS:
Overall Officials: SANDRINE MESTRE, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - CHU Montpellier - Hôpital St Eloi - Service Maladies Vasculaires, Montpellier
  - Hôpital Cognacq-Jay - unité de lymphologie, Paris
  - CHU TOULOUSE - service médecine vasculaire, Toulouse

REFERENCES:
- [Background] Garaffa G, Christopher N, Ralph DJ. The management of genital lymphoedema. BJU Int. 2008 Aug;102(4):480-4. doi: 10.1111/j.1464-410X.2008.07559.x. Epub 2008 Mar 5. PMID 18325055
- [Background] Facio MF, Spessoto LC, Gatti M, Ferraz Arruda PF, Ferraz Arruda JG, Antoniassi TS, Bogdan AP, Godoy MF, Godoy JM, Facio FN Jr. Clinical Treatment of Penile Fibrosis After Penoscrotal Lymphedema. Urol Case Rep. 2017 Jan 5;11:14-16. doi: 10.1016/j.eucr.2016.12.001. eCollection 2017 Feb. PMID 28083477
- [Background] Shim TN, Doiron PR, Francis N, Minhas S, Muneer A, Hawkins D, Dinneen M, Bunker CB. Penile lymphoedema: approach to investigation and management. Clin Exp Dermatol. 2019 Jan;44(1):20-31. doi: 10.1111/ced.13609. Epub 2018 Jul 15. PMID 30009576
- [Derived] Mestre S, Vignes S, Malloizel-Delaunay J, Abba S, Villet S, Picolet A, Vicaut E, Quere I. Positive Impact of a New Compressive Garment in Patients with Genital Lymphedema: OLYMPY Study. Lymphat Res Biol. 2024 Apr;22(2):138-146. doi: 10.1089/lrb.2023.0055. Epub 2024 Apr 2. PMID 38563697